CLINICAL TRIAL: NCT03692858
Title: IPACK Block Efficacy as a Part of Multimodal Analgesia in Total Knee Arthroplasty. A Prospective, Randomized, Controlled, Double Blinded Study
Brief Title: IPACK Block in Total Knee Arthroplasty
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asklepieion Voulas General Hospital (Other Government)
Collaborators: Aikaterini Kalampokini (Unknown); Chryssoula Staikou (Unknown)
Responsible Party: Principal Investigator, Alexandros Makris, Consultant Anesthesiologist, Asklepieion Voulas General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8885/20-06-2018
Record Dates: First submitted 2018-09-30; First posted 2018-10-02 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Total Knee Arthroplasty
Keywords: arthroplasty; replacement; knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator)
  Interventions: Drug: Adductor Canal Block plus IPACK Block
- Group B (Active Comparator)
  Interventions: Drug: Adductor Canal Block

INTERVENTIONS:
Drug: Adductor Canal Block plus IPACK Block — Adductor Canal Block plus IPACK Block using Ropivacaine
  Arms: Group A
Drug: Adductor Canal Block — Adductor Canal Block using Ropivacaine
  Arms: Group B

SUMMARY:
100 patients ASA I-III, undergoing total knee arthroplasty under spinal anesthesia, will be randomly assigned into one of two groups, namely group A (n=50), where an adductor canal block and an IPACK block will be performed preoperatively and group B (n=50) where an adductor canal block only will be performed preoperatively. All patients will receive a standardized multimodal approach, including pregabalin, paracetamol, and PCA with morphine. NRS scores in static and dynamic conditions during the first 48 hours postoperatively, morphine consumption during the first 24 hours postoperatively will be measured and additionally, patient satisfaction, complications, range of knee motion, moblization, functionality, delirium ocurence will be recorded. Chronic pain will be assessed in 3 and 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Physical status according to American Society of Anesthesiologists (ASA) I-III
* Patients scheduled for total knee arthroplasty

Exclusion Criteria:

* Previous operation on same knee
* Contraindication of spinal anesthesia, peripheral nerve blocks or any of the agents used in the protocol
* BMI above 32
* Serious psychiatric, mental and cognitive disorders
* Language barrier
* Block failure
* Chronic opioid, gabapentinoid use
* Severe kidney disfunction

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
NRS scores | 48 hours
  Numerical Rating Scale (NRS) scores (Range 0-10, 0=no pain, 10=the worse pain ever)
Morphine consumption | 24 hours
  Morphine consumption in mg
Chronic pain | 6 months
  Using of Graded Chronic Pain Scale (GCPS) Grade 0: No pain in prior 6 months Grade 1: Low Intensity - Low Disability Grade II: High Intensity Characteristic Pain Intensity - Low Disability Grade III: High Disability - Moderately Limiting Grade IV: High Disability - Severely Limiting

SECONDARY OUTCOMES:
Delirium occurence | 48 hours
  Nu-DESK scale (presence of disorientation, inappropriate behavior, inappropriate communication,illusions/hallucinations, psychomoter retardation). Each of the 5 items is rated from 0 to 2. A total of 10 is the maximum score. A score of more than 2 identifies the presence of delirium.
Range of knee motion | 48 hours
  Degrees of flexion
Complications | 48 hours
Patient mobilization | 5 days
  Patient reporting time of first standing to the side of the bed and number of steps per day
Patient satisfaction | 48 hours
  Patients asked whether they would choose the same anaesthetic management in a future operation: Yes/No
Joint function | 6 months
  Maximal flexion / extension
Intestinal function | 5 days
  Time of first passing of rectal gas, reported by the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Asklepieion Hospital of Voula, Athens, Greece